CLINICAL TRIAL: NCT00305682
Title: Transplantation of Unrelated Donor Umbilical Cord Blood in Patients With Hematological Malignancies Using a Non-Myeloablative Preparative Regimen
Brief Title: Non-Myeloablative Conditioning for Unrelated Donor Umbilical Cord Blood Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS036; UMN-MT-2005-02 (Other: Blood and Marrow Transplantation Program); UMN-0507M70121 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1-Previous Autologous Transplant (Active Comparator): Arm 1 - hematologic malignancy patients who have received a previous autologous transplant or ≥ 2 cycle of multiagent chemotherapy within the last 3 months previous to umbilical cord blood transplant (UCBT). Conditioning Fludarabine dose of 40 mg/m2/day x 5, cyclophosphamide and total body irradiation without anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus
- Arm 2 - No Prior Autologous Transplant (Active Comparator): Arm 2 - hematologic malignancy patients who have not been treated with prior autologous transplant or ≤ 1 cycle of chemotherapy in the 3 months previous to umbilical cord blood transplant (UCBT), and who should receive anti-thymocyte globulin as conditioning regimen. Conditioning Fludarabine dose of 40 mg/m2/day x 5, cyclophosphamide and total body irradiation with anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus
- Arm 3 - Refractory Leukemia/Lymphoma (Active Comparator): Arm 3 - patients with refractory leukemia or lymphoma who have been rendered aplastic either by induction chemotherapy or radioimmunoconjugated monoclonal antibody therapy. Conditioning Fludarabine dose of 40 mg/m2/day x 5, cyclophosphamide and total body irradiation with anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus
- Arm 4: MT2006-01 coenrolling patients (Active Comparator): Arm 4 - hematologic malignancy patients enrolled in MT2006-01. Conditioning Fludarabine dose of 40 mg/m2/day x 5, cyclophosphamide and total body irradiation with or without anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus
- Arm 5 - Previous Autologous Transplant (Active Comparator): Arm 5 - hematologic malignancy patients who have received a previous autologous transplant or ≥ 2 cycle of multiagent chemotherapy within the last 3 months previous to umbilical cord blood transplant (UCBT). Conditioning Fludarabine dose of 30 mg/m2/day x 5, cyclophosphamide and total body irradiation without anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus
- Arm 6 - No prior autologous transplant (Active Comparator): Arm 6 - hematologic malignancy patients who have not been treated with prior autologous transplant or ≤ 1 cycle of chemotherapy in the 3 months previous to umbilical cord blood transplant (UCBT), and who should receive anti-thymocyte globulin as conditioning regimen. Conditioning Fludarabine dose of 30 mg/m2/day x 5, cyclophosphamide and total body irradiation with anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: Fludarabine; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total body irradiation; Drug: Sirolimus

INTERVENTIONS:
Biological: anti-thymocyte globulin — Equine ATG dose is 15 mg/kg intravenously (IV) every 12 hours for 6 doses on days -6, - 5, and -4.
  Other Names: ATGAM; ATG
  Arms: Arm 2 - No Prior Autologous Transplant; Arm 3 - Refractory Leukemia/Lymphoma; Arm 6 - No prior autologous transplant
Drug: cyclophosphamide — Cyclophosphamide 50mg/kg x 1 to be administered IV over 2 hours with high volume fluid flush on day -6.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine 40 mg/m2/day or 30 mg/m2/day intravenously (IV) as one hour infusion x 5 days, on day -6 to -2.
  Other Names: Fludara
Drug: mycophenolate mofetil — Mycophenolate mofetil (MMF) 3 gram/day for patients who are ≥ 40 kg divided in 2 or 3 doses. Pediatric patient (<40 kilograms) will receive MMF at the dose of 15 mg/kg/dose every 8 hours.
  Other Names: MMF
Procedure: umbilical cord blood transplantation — One or 2 UCB units may be infused to achieve the required cell dose.
  Other Names: UCBT
Radiation: total body irradiation — Administered Day -1, 200 cGy
  Other Names: TBI
Drug: Sirolimus — Sirolimus will be administered starting at day -3 with 8mg-12mg mg oral loading dose followed by single dose 4 mg/day with a target serum concentration of 3 to 12 mg/mL. Levels are to be monitored 3 times/week in the first 2 weeks, weekly until day +60, and as clinically indicated until day +100 post-transplantation. In the absence of acute GVHD sirolimus may be tapered starting at day +100 and eliminated by day +180 post-transplantation.
  Other Names: rapamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. An umbilical cord blood transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving sirolimus and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation followed by an umbilical cord blood transplant, sirolimus, and mycophenolate mofetil works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the one- and two-year survival of patients with hematologic malignancies treated with a nonmyeloablative conditioning regimen comprising fludarabine, cyclophosphamide, and total-body irradiation followed by umbilical cord blood transplantation and post-transplant immunosuppression comprising sirolimus and mycophenolate mofetil.

Secondary

* Determine the six-month nonrelapse mortality of patients treated with this regimen.
* Determine the presence of chimerism in patients treated with this regimen at days 21, 60, 100, 180, and 365.
* Determine the incidence of neutrophil engraftment by day 42 in patients treated with this regimen.
* Determine the incidence of platelet engraftment by six months in patients treated with this regimen.
* Determine the incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) at day 100 in patients treated with this regimen.
* Determine the incidence of chronic GVHD at one year in patients treated with this regimen.
* Determine the probability of overall survival within one or two years in patients treated with this regimen.
* Determine the probability of progression-free survival within one or two years in patients treated with this regimen.
* Determine the incidence of relapse or disease progression within one or two years in patients treated with this regimen.

OUTLINE: This is a nonrandomized study. Patients are stratified into five disease groups: 1. acute myeloid leukemia, myelodysplastic syndromes, chronic myelogenous leukemia [CML] in first chronic phase and second chronic phase [CP2] after myeloid blast crisis; 2. acute lymphoblastic leukemia, Burkitt's lymphoma, CML CP2 post lymphoid blast crisis, 3. large-cell B and T-cell lymphoma, mantle cell lymphoma; 4. chronic lymphocytic leukemia/small lymphocytic lymphoma, prolymphocytic leukemia, marginal zone B-cell lymphoma, follicular lymphoma; 5. Hodgkin's lymphoma and multiple myeloma.

* Nonmyeloablative conditioning: Patients receive fludarabine intravenously on days -6 to -2 and cyclophosphamide IV on day -6. Patients who did not undergo prior autologous transplant or who received ≤ 1 course of prior multiagent chemotherapy or no severely immunosuppressive therapy in the past 3 months also receive anti-thymocyte globulin IV on days -6 to -4. All patients also undergo total-body irradiation on day -1.
* Umbilical cord blood transplant: Patients undergo umbilical cord blood transplantation on day 0.
* Post-transplant immunosuppression: Sirolimus will be administered starting at day -3 with 8mg-12mg mg oral loading dose followed by single dose 4 mg/day with a target serum concentration of 3 to 12 mg/mL. Levels are to be monitored 3 times/week in the first 2 weeks, weekly until day +60, and as clinically indicated until day +100 post-transplantation. In the absence of acute GVHD sirolimus may be tapered starting at day +100 and eliminated by day +180 post-transplantation. Patients also receive mycophenolate mofetil IV on days -3 to 5 and then orally on days 6-30.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 320 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

Age, Graft Cell Dose and Graft HLA Criteria

* Subjects must be <70 years old. Subjects ages ≥ 70 and ≤ 75 may be eligible if they have a Co-Morbidity Scoring (HCT-CI) score ≤ 2.
* The UCB graft is matched at 4-6 HLA-A, B, DRB1 antigens with the recipient.
* Patients co-enrolled in MT-2006-01 Phase I Study of Infusion of Umbilical Cord Blood Derived CD25+CD4+ T-Regulatory (Treg) Cells after Non-Myeloablative Cord\Blood Transplantation will receive grafts composed of 2 UCB units.

Disease Criteria:

* Acute Leukemias:

  * Acute myeloid leukemia: high risk complete remission 1 (CR1) (as evidenced by preceding myelodysplastic syndrome (MDS), high risk cytogenetics such as those associated with MDS or complex karyotype, > 2 cycles to obtain CR or erythroblastic and megakaryocytic); second or greater CR.
  * Acute lymphoblastic leukemia/lymphoma: high risk CR1 as evidenced by high risk cytogenetics (e.g. t(9;22), t(1;19),t(4;11), other myeloid/lymphoid or mixed lineage leukemia [MLL] rearrangements, hypodiploidy or Ikaros family zinc finger 1 [IKZF1]), > 1 cycle to obtain CR or evidence of minimal residual disease (MRD). Patients in second or greater CR are also eligible.
* Burkitt's lymphoma in CR2 or subsequent CR
* Natural Killer cell malignancies
* Chronic myelogenous leukemia: all types except refractory blast crisis. Chronic phase patients must have failed or been intolerant to Gleevec
* Myelodysplastic syndrome:
* Large-cell lymphoma, Hodgkin lymphoma and multiple myeloma with chemotherapy sensitive disease that has failed or patients who are ineligible for an autologous transplant.
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma, which have progressed within 12 months of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease should be considered for debulking chemotherapy before transplant. Patients with refractory disease are eligible, unless has bulky disease and an estimated tumor doubling time of less than one month.
* Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy if chemotherapy sensitive.
* Refractory leukemia or MDS.
* Bone marrow failure syndromes, except for Fanconi Anemia
* Myeloproliferative syndromes Patients who have undergone an autologous transplant >12 months prior to allogeneic transplantation

Adequate Organ Function and Performance Status

Exclusion Criteria:

* < 70 years with an available 5-6/6 HLA-A, B, DRB1 matched sibling donor
* Pregnancy or breastfeeding
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Current active serious infection
* Unless in post-chemotherapy and radioimmunoconjugated antibody induced aplasia, when he/she would be eligible for Arm 3, patients with acute leukemia in morphologic relapse/ persistent disease defined as > 5% blasts in normocellular bone marrow OR any % blasts if blasts have unique morphologic markers (e.g. Auer rods) or associated cytogenetic markers that allows morphologic relapse to be distinguished are not eligible.
* Chronic myelogenous leukemia (CML) in refractory blast crisis
* Large cell lymphoma, mantle cell lymphoma and Hodgkin disease that is progressive on salvage therapy. Stable disease is acceptable to move forward provided it is non-bulky.
* Active central nervous system malignancy

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Bachanova V, Verneris MR, DeFor T, Brunstein CG, Weisdorf DJ. Prolonged survival in adults with acute lymphoblastic leukemia after reduced-intensity conditioning with cord blood or sibling donor transplantation. Blood. 2009 Mar 26;113(13):2902-5. doi: 10.1182/blood-2008-10-184093. Epub 2009 Jan 28. PMID 19179301
- [Result] Brunstein CG, Cantero S, Cao Q, Majhail N, McClune B, Burns LJ, Tomblyn M, Miller JS, Blazar BR, McGlave PB, Weisdorf DJ, Wagner JE. Promising progression-free survival for patients low and intermediate grade lymphoid malignancies after nonmyeloablative umbilical cord blood transplantation. Biol Blood Marrow Transplant. 2009 Feb;15(2):214-22. doi: 10.1016/j.bbmt.2008.11.013. PMID 19167681
- [Derived] Bachanova V, Burke MJ, Yohe S, Cao Q, Sandhu K, Singleton TP, Brunstein CG, Wagner JE, Verneris MR, Weisdorf DJ. Unrelated cord blood transplantation in adult and pediatric acute lymphoblastic leukemia: effect of minimal residual disease on relapse and survival. Biol Blood Marrow Transplant. 2012 Jun;18(6):963-8. doi: 10.1016/j.bbmt.2012.02.012. Epub 2012 Mar 16. PMID 22430088
- [Derived] Bachanova V, Sandhu K, Yohe S, Cao Q, Burke MJ, Verneris MR, Weisdorf D. Allogeneic hematopoietic stem cell transplantation overcomes the adverse prognostic impact of CD20 expression in acute lymphoblastic leukemia. Blood. 2011 May 12;117(19):5261-3. doi: 10.1182/blood-2011-01-329573. Epub 2011 Mar 14. PMID 21403127
- [Derived] MacMillan ML, Weisdorf DJ, Brunstein CG, Cao Q, DeFor TE, Verneris MR, Blazar BR, Wagner JE. Acute graft-versus-host disease after unrelated donor umbilical cord blood transplantation: analysis of risk factors. Blood. 2009 Mar 12;113(11):2410-5. doi: 10.1182/blood-2008-07-163238. Epub 2008 Nov 7. PMID 18997171
- See also: https://pubmed.ncbi.nlm.nih.gov/19179301/ — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4582655/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 patients were excluded from receiving the treatment as they were not eligible. 4 patients were removed from the study because the participating site withdrew the participation from the study
Groups:
- Arm 1-Previous Autologous Transplant: hematologic malignancy patients who have received a previous autologous transplant or ≥ 2 cycle of multiagent chemotherapy within the last 3 months previous to umbilical cord blood transplant (UCBT). Conditioning Fludarabine dose of 40 mg/m2/day x 5, cyclophosphamide and total body irradiation without anti-thymocyte globulin followed by umbilical cord blood transplantation, and peri-transplant Mycophenolate Mofetil and Sirolimus.
Period: Overall Study
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Started | 98 | 71 | 7 | 34 | 39 | 35
Completed | 98 | 71 | 7 | 34 | 39 | 35
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant | Total
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 0 | 0 | 0 | 1 | 11
  Between 18 and 65 years | 79 | 55 | 6 | 30 | 29 | 19 | 218
  >=65 years | 12 | 13 | 1 | 4 | 10 | 15 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 5 | 16 | 14 | 15 | 116
  Male | 61 | 42 | 2 | 18 | 25 | 20 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 1 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 6 | 1 | 0 | 2 | 0 | 1 | 10
  White | 82 | 61 | 5 | 31 | 39 | 30 | 248
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 9 | 4 | 1 | 0 | 0 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 98 | 71 | 7 | 34 | 39 | 35 | 284

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Alive at 1 Year Post Transplant
Description: Overall Survival - Number of patients alive at 1 year post transplant
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 59 | 40 | 1 | 26 | 26 | 25

2. Primary Outcome: Number of Participants Who Were Alive at 2 Years Post Transplant
Description: Overall Survival - Number of patients alive at 2 years post transplant
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 50 | 31 | 1 | 20 | 21 | 23

3. Secondary Outcome: Number of Participants Who Were Dead at 6 Months After Study Completion
Description: Incidence of Non-relapse mortality - Number of Patients Dead at 6 Months after study completion
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 10 | 20 | 2 | 5 | 3 | 6

4. Secondary Outcome: Percentage of Donor Chimerism at 21 Days
Description: Chimerism studies will be performed on the blood and bone marrow (BM). BM chimerism days 21 and 100, at 6 months and 1 year to determine the relative contribution of donor and recipient hematopoiesis.
Time Frame: 21 days
Population: A total of 43 participants were not evaluable
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 86 | 61 | 6 | 25 | 35 | 28
percentage of donor cells | 77 (25) | 73 (32) | 57 (29) | 77 (21) | 69 (32) | 68 (33)

5. Secondary Outcome: Percentage of Donor Chimerism at 100 Days
Description: as for outcome 4
Time Frame: 100 days
Population: A total of 85 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 64 | 50 | 2 | 30 | 27 | 26
percentage of donor cells | 94 (18) | 94 (21) | 100 (0) | 93 (23) | 85 (31) | 86 (32)

6. Secondary Outcome: Percentage of Donor Chimerism at 180 Days
Description: as for outcome 4
Time Frame: 180 Days
Population: A total of 134 participants were not evaluable
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 49 | 32 | 2 | 22 | 22 | 23
percentage of donor cells | 96 (18) | 98 (6) | 88 (17) | 94 (16) | 91 (26) | 98 (10)

7. Secondary Outcome: Percentage of Donor Chimerism at 365 Days
Description: as for outcome 4
Time Frame: 365 days
Population: A total of 160 participants were not evaluable
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 42 | 27 | 0 | 19 | 16 | 20
percentage of donor cells | 99 (2) | 98 (12) |  | 99 (6) | 87 (34) | 100 (0)

8. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Time to 1st 3 consecutive days with absolute neutrophil count (ANC) > 5 x 10^8/L and percentage of patients with neutrophil recovery by day 42 (Cumulative incidence).
Time Frame: Day 42
Population: 7 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 97 | 67 | 7 | 34 | 38 | 34
Participants | 93 | 65 | 6 | 32 | 32 | 29

9. Secondary Outcome: Number of Participants With Platelet Engraftment
Description: Time to platelets > 20,000 (first of 3 consecutive days) with no platelet transfusions for seven days and percentage of patients with platelet engraftment >50,000 by day 100.
Time Frame: Day 180
Population: 13 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 96 | 63 | 7 | 34 | 37 | 34
Participants | 75 | 47 | 3 | 28 | 34 | 25

10. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD)
Description: Determine the incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) at day 100 post transplant. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria used for staging.
  Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 45 | 24 | 1 | 12 | 13 | 13

11. Secondary Outcome: Number of Participants With Chronic Graft-Versus-Host Disease
Description: Determine the incidence of chronic GVHD at 1 year after transplant. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 18 | 20 | 0 | 3 | 3 | 3

12. Secondary Outcome: Number of Participants Experiencing Progression-free Survival
Description: Incidence of Progression-free survival - Number of patients who were alive and did not have disease progression. Patients with leukemia and lymphoma involving the bone marrow (BM) and multiple myeloma will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients with lymphoma and myeloma will have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 43 | 32 | 1 | 21 | 16 | 24

13. Secondary Outcome: Number of Participants Experiencing Progression-free Survival at 2 Years
Description: Incidence of Progression-free survival - Number of patients who were alive and did not have disease progression
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 36 | 25 | 1 | 17 | 16 | 20

14. Secondary Outcome: Number of Participants Experiencing Relapse (Incidence of Relapse)
Description: Patients with leukemia and lymphoma involving the BM and multiple myeloma will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients with lymphoma and myeloma will have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 43 | 14 | 4 | 7 | 20 | 2

15. Secondary Outcome: Number of Participants Experiencing Relapse (Incidence of Relapse) at 2 Years
Description: as for outcome 14
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
Number analyzed (Participants) | 98 | 71 | 7 | 34 | 39 | 35
Participants | 49 | 19 | 4 | 11 | 20 | 4

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm 1-Previous Autologous Transplant | Arm 2 - No Prior Autologous Transplant | Arm 3 - Refractory Leukemia/Lymphoma | Arm 4: MT2006-01 Coenrolling Patients | Arm 5 - Previous Autologous Transplant | Arm 6 - No Prior Autologous Transplant
All-Cause Mortality (participants affected / at risk) | 48/98 | 40/71 | 6/7 | 14/34 | 18/39 | 12/35
Serious Adverse Events (participants affected / at risk) | 53/98 | 48/71 | 3/7 | 11/34 | 2/39 | 4/35
Other Adverse Events (participants affected / at risk) | 76/98 | 54/71 | 5/7 | 20/34 | 33/39 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Previous Autologous Transplant (N=98) | Arm 2 - No Prior Autologous Transplant (N=71) | Arm 3 - Refractory Leukemia/Lymphoma (N=7) | Arm 4: MT2006-01 Coenrolling Patients (N=34) | Arm 5 - Previous Autologous Transplant (N=39) | Arm 6 - No Prior Autologous Transplant (N=35)
Graft versus host disease (Immune system disorders) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Primary Graft Failure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood/Bone Marrow,other - relapse disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Bone marrow cellularity - aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular, other disorder - substernal chest discomfort (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CNS hemorrhage/bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 24 (24) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 11 (11) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Leukoencephalopathy associated with radiological findings (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillamme Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Previous Autologous Transplant (N=98) | Arm 2 - No Prior Autologous Transplant (N=71) | Arm 3 - Refractory Leukemia/Lymphoma (N=7) | Arm 4: MT2006-01 Coenrolling Patients (N=34) | Arm 5 - Previous Autologous Transplant (N=39) | Arm 6 - No Prior Autologous Transplant (N=35)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8 (16) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 8 (9) | 6 (6) | 1 (1) | 1 (1) | 4 (7) | 2 (3)
Cytomegaloviral infection (Infections and infestations) | 13 (14) | 5 (6) | 1 (2) | 2 (2) | 1 (1) | 6 (6)
Dialysis (Renal and urinary disorders) | 4 (4) | 8 (9) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Deep vein thrombosis (DVT) (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Engraftment syndrome (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 7 (7) | 3 (3)
GI disorder (Gastrointestinal disorders) | 5 (6) | 3 (4) | 0 (0) | 2 (3) | 3 (3) | 3 (3)
Heart disorder (Cardiac disorders) | 4 (7) | 6 (10) | 1 (1) | 3 (4) | 6 (10) | 7 (10)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 5 (5)
hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 9 (9) | 10 (10)
Infection (Infections and infestations) | 32 (114) | 18 (51) | 4 (23) | 11 (27) | 33 (101) | 33 (122)
Intubation (Respiratory, thoracic and mediastinal disorders) | 12 (20) | 15 (20) | 2 (5) | 5 (7) | 2 (2) | 6 (10)
mastoiditis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neuropathy (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 3 (3)
neurotoxicity (Nervous system disorders) | 2 (3) | 11 (14) | 2 (4) | 1 (1) | 2 (3) | 3 (4)
pericardial effusion (Cardiac disorders) | 10 (11) | 14 (17) | 1 (1) | 4 (4) | 5 (6) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 39 (86) | 37 (81) | 4 (15) | 13 (28) | 18 (37) | 20 (60)
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (11) | 3 (3) | 1 (1) | 1 (1) | 4 (5)
Seizure (Nervous system disorders) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Skin rashes due to drug toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (3) | 1 (1)
Supraventricular tachycardia (SVT) (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT00305682/Prot_SAP_000.pdf